CLINICAL TRIAL: NCT02402088
Title: The Purpose of This Study is to Investigate the Role of Stress in Food Craving and Food Consumption by Examining Stress Response Using Subjective, Physiological and Neurobiological Measurements
Brief Title: The Role of Emotional Arousal in Food Preference and Taste
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 0801003403; 1R01DK099039-01A1 (NIH)
Record Dates: First submitted 2014-01-30; First posted 2015-03-30 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Obesity; Food Craving; Food Consumption
Keywords: stress; food cues; obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Normal Weight (Active Comparator): BMI18.5-24.9 (normal range)
  Interventions: Behavioral: Stress Imagery; Behavioral: Food Cue Imagery; Behavioral: Neutral-Relaxing
- Overweight (Experimental): body mass index between 25.0 - 29.9 (overweight range)
  Interventions: Behavioral: Stress Imagery; Behavioral: Food Cue Imagery; Behavioral: Neutral-Relaxing
- Obese (Experimental): body mass index between 30 and 35 (obese range)
  Interventions: Behavioral: Stress Imagery; Behavioral: Food Cue Imagery; Behavioral: Neutral-Relaxing

INTERVENTIONS:
Behavioral: Stress Imagery — The stress imagery script will be based on subjects' description of a recent personal stressful event that they had experienced as "most stressful". "Most stressful" is determined by having the subjects rate the perceived stress experienced by them on a 10-point Likert scale where "1=not at all stressful" and "10=the most stress they felt recently in their life". Only situations rated as 8 or above on this scale are accepted as appropriate for script development. Examples of acceptable stressful situations include breakup with significant other, a verbal argument with a significant other or family member or unemployment-related stress, such as being fired or laid off from work.
Behavioral: Food Cue Imagery — A food cue script will be developed from the subjects' experience of eating their most favorite foods. Examples include ordering pizza, cooking a favorite meal, or going out to a restaurant.
Behavioral: Neutral-Relaxing — A neutral-relaxing script will be developed from the subjects' commonly experienced neutral-relaxing situations, such as a trip to the beach or park.

SUMMARY:
The purpose of this study is to examine the role of stress in food craving and food consumption in obesity. Using experimentally validated guided imagery procedure, the investigators propose to examine the stress response using subjective, physiological and neurobiological measurements.

DETAILED DESCRIPTION:
One hundred and fifty men and women will participate in three laboratory sessions to assess stress responses to personal stress imagery, food cue imagery, and to neutral-relaxing imagery. Subjects will be distributed into 3 groups stratified by BMI category. Subject recruitment, eligibility determination, baseline assessments and script development will be conducted at the Yale Stress Center. Subjects will complete a variety of diagnostic, cognitive and psychological assessments, a comprehensive physical examination and blood work and will be involved in development of imagery scripts from personal stress, food cue and neutral-relaxing situations. Subjects will then be scheduled for three laboratory sessions at the Yale Stress Center. Subjects will also participate in an imagery and relaxation training session followed by three laboratory sessions. The three laboratory sessions will be conducted within a brief interval of days, when subjects will be exposed to a personal stress, a food cue and a neutral-relaxing imagery condition, one condition per day. The order of imagery conditions will be randomly assigned and counterbalanced across subjects in order to balance any influences due to order of imagery conditions.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 18-45 years
* Able to read and write
* Normal/lean BMI group: BMI 18.5-24.9 as calculated based on height and weight.
* Overweight BMI group: BMI 25.0 - 29.9 as calculated based on height and weight Obese BMI group: BMI 30-35 as calculated based on height and weight.
* Do not meet criteria for any current Axis I DSM-IV psychiatric diagnoses and provide negative urine toxicology screens during initial appointments and at admission for laboratory sessions.

Exclusion Criteria:

* Meet current criteria for dependence on any psychoactive substance, including nicotine and caffeine
* Current use of any psychoactive drugs, including anxiolytics, antidepressants, naltrexone or antabuse
* Any psychotic disorder or current psychiatric symptoms requiring specific attention, including need for psychiatric medications for current major depression and anxiety disorders
* Any significant current medical condition such as neurological, cardiovascular, endocrine, renal, liver, thyroid pathology; subjects on medications for any medical condition will be excluded
* Women on oral contraceptives, peri and post menopausal women, and those with hysterectomies
* Pregnant and lactating women will be excluded.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Food Craving based on the Food Craving Inventory | Baseline
  An abbreviated assessment base don the Food Craving Inventory. The Food Craving Inventory is a self-report questionnaire of specific food cravings. The questionnaire consists of 25 items measuring the frequency of cravings for specific foods and consists of 4 factors or subscales measuring cravings for High Fats, Carbohydrates/Starches, Sweets, and Fast Food Fats and also generates a total score. The brief version of the inventory uses 2 items from each of the 4 subscales.
Food Craving based on the Food Craving Inventory | Immediately After Image
  An abbreviated assessment base don the Food Craving Inventory. The Food Craving Inventory is a self-report questionnaire of specific food cravings. The questionnaire consists of 25 items measuring the frequency of cravings for specific foods and consists of 4 factors or subscales measuring cravings for High Fats, Carbohydrates/Starches, Sweets, and Fast Food Fats and also generates a total score. The brief version of the inventory uses 2 items from each of the 4 subscales.
Food Craving based on the Food Craving Inventory | 5 minutes
  An abbreviated assessment base don the Food Craving Inventory at plus 5 minutes. The Food Craving Inventory is a self-report questionnaire of specific food cravings. The questionnaire consists of 25 items measuring the frequency of cravings for specific foods and consists of 4 factors or subscales measuring cravings for High Fats, Carbohydrates/Starches, Sweets, and Fast Food Fats and also generates a total score. The brief version of the inventory uses 2 items from each of the 4 subscales.
Food Craving based on the Food Craving Inventory | 15 minutes
  An abbreviated assessment base don the Food Craving Inventory at plus 15 minutes. The Food Craving Inventory is a self-report questionnaire of specific food cravings. The questionnaire consists of 25 items measuring the frequency of cravings for specific foods and consists of 4 factors or subscales measuring cravings for High Fats, Carbohydrates/Starches, Sweets, and Fast Food Fats and also generates a total score. The brief version of the inventory uses 2 items from each of the 4 subscales.
Food Craving based on the Food Craving Inventory | 30 minutes
  An abbreviated assessment base don the Food Craving Inventory at plus 30 minutes. The Food Craving Inventory is a self-report questionnaire of specific food cravings. The questionnaire consists of 25 items measuring the frequency of cravings for specific foods and consists of 4 factors or subscales measuring cravings for High Fats, Carbohydrates/Starches, Sweets, and Fast Food Fats and also generates a total score. The brief version of the inventory uses 2 items from each of the 4 subscales.
Food Craving based on the Food Craving Inventory | 45 minutes
  An abbreviated assessment base don the Food Craving Inventory at plus 45 minutes. The Food Craving Inventory is a self-report questionnaire of specific food cravings. The questionnaire consists of 25 items measuring the frequency of cravings for specific foods and consists of 4 factors or subscales measuring cravings for High Fats, Carbohydrates/Starches, Sweets, and Fast Food Fats and also generates a total score. The brief version of the inventory uses 2 items from each of the 4 subscales.
Food Craving based on the Food Craving Inventory | 60 minutes
  An abbreviated assessment base don the Food Craving Inventory at plus 60 minutes. The Food Craving Inventory is a self-report questionnaire of specific food cravings. The questionnaire consists of 25 items measuring the frequency of cravings for specific foods and consists of 4 factors or subscales measuring cravings for High Fats, Carbohydrates/Starches, Sweets, and Fast Food Fats and also generates a total score. The brief version of the inventory uses 2 items from each of the 4 subscales.

SECONDARY OUTCOMES:
food snack intake | 30 minutes
  Food snacks are offered after each imagery condition and weighed for snack consumption.After each imagery period, subjects are presented with 3 bowls of highly palatable (chocolate pudding; potato chips, mini chocolate chip cookies) and 3 bowls of healthy food snacks (baby carrots; grapes), each portioned to ~500 calories (3000 calories per lab session).

CONTACTS AND LOCATIONS:
Overall Officials: Rajita Sinha, PhD, Principal Investigator — Professor
Locations (1):
- Yale University, New Haven, Connecticut, United States